CLINICAL TRIAL: NCT03200314
Title: Measurment of Blood Recirculation and Adjustment of vvECMO Blood Flow During Veno-venous Extracoporeal Membrane Oxygenation
Brief Title: Blood Recirculation and vvECMO
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Steffen Weber-Carstens, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: EA208317
Record Dates: First submitted 2017-06-26; First posted 2017-06-27 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: ARDS; Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measurment of blood recirculation — Ultrasound based measurments of blood recirculating through the vvECMO circuit.

SUMMARY:
A prospective, observational study will be performed measuring recirculation of blood through a veno-venous Extracoporeal Membrane Oxygenation (vvECMO) in patients with acute respiratory distress syndrome (ARDS) on vvECMO. ECMO blood flow will be adjusted with respect to recirculation.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or older
* ARDS
* veno-venous ECMO

Exclusion Criteria:

* age < 18 years
* hemodynamic instability during measurement of recirculation
* pregnancy
* inability to obtain patient's consent or consent of legal guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older requiring veno-venous ECMO for treatment of refractory hypomxemia in ARDS.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2017-08-13 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
Recirculation of vvECMO blood flow | Once within first week after ICU admission during 4 hours
  Amount of ECMO blood flow recirculating through the vvECMO circuit

SECONDARY OUTCOMES:
Reduction of vvECMO blood flow | Once within first week after ICU admission during 4 hours
  Reduction of vvECMO blood flow if a significant recirculation can be measured
Arterial blood oxygen content after reduction of vvECMO blood flow | Once within first week after ICU admission during 4 hours
  Change in arterial blood oygen content after reduction of vvECMO blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Martin Russ, Dr. med., Principal Investigator — Charite University Hospital Berlin; Philipp A Pickerodt, Dr. med., Principal Investigator — Charite University Hospital Berlin; Steffen Weber-Carstens, PD Dr. med., Principal Investigator — Charite University Hospital Berlin
Locations (1):
- Charite University, Berlin, Germany, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No